CLINICAL TRIAL: NCT00529776
Title: Prophylaxis of Ventilator Associated Pneumonia by Continuous Lateral Rotation Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Thomas Staudinger, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: EK 38/2004
Record Dates: First submitted 2007-09-12; First posted 2007-09-14 (Estimated); Last update posted 2008-06-11 (Estimated); Status verified 2008-06

CONDITIONS: Pneumonia, Ventilator-Associated
Keywords: Prevention of ventilator associated pneumonia
MeSH Terms: conditions — Pneumonia, Ventilator-Associated

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Continuous lateral rotation therapy
  Interventions: Procedure: Continuous lateral rotation therapy
- 2 (No Intervention): Standard manual positioning (Supine position)

INTERVENTIONS:
Procedure: Continuous lateral rotation therapy
  Arms: 1

SUMMARY:
Hypothesis: Ventilator associated pneumonia (VAP) in critically ill patients may be prevented by continuous lateral rotation therapy (CLRT) using specially designed, motor driven beds.

Patients are randomized to CLRT or supine position if mechanically ventilated and not suffering from pneumonia or ARDS within 48 hours after intubation. Prophylaxis of VAP is standardized in both groups. Primary endpoint is incidence of VAP, secondary endpoints are length of ventilation, length of stay and mortality.

ELIGIBILITY:
Inclusion Criteria:

* Mechanically ventilated
* Intubated not longer than 48 h
* Medical cause for ICU admission
* Expected to be ventilated for > 48 hours

Exclusion Criteria:

* Pneumonia or ARDS present
* Postoperative patient

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2005-09; Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Ventilator associated pneumonia

SECONDARY OUTCOMES:
Length of hospital stay
Length of mechanical ventilation
ICU and hospital Mortality

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Staudinger, MD, Principal Investigator — Department of Internal Medicine I, Medical University of Vienna, Austria; Thomas Staudinger, MD, Principal Investigator — Dept. of Internal Medicine I, Medical University of Vienna
Locations (1):
- Vienna General Hospital, Medical University of Vienna, Vienna, Austria